CLINICAL TRIAL: NCT03635541
Title: Dynamic Changes and Risk Factors of Fibrosis and Steatosis Progression in Nonalcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hong You, Vice-Director of Liver Research Center, Beijing Friendship Hospital
Other Study IDs: YYYY-2018-NAFLD
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: non alcoholic fatty liver disease; non alcoholic steatohepatitis; steatosis; fibrosis; progression; risk factors
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Fibrosis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational group of NAFLD: Liver biopsy proved NAFLD patients, observational study. Oral advice on lifestyle would be given at each visit.
  Interventions: Other: observational group of NAFLD

INTERVENTIONS:
Other: observational group of NAFLD — there's no intervention for patients for it is a observational study

SUMMARY:
It is an observational study of non alcoholic fatty liver disease (NAFLD) patients with a calculated sample size of 90. Liver biopsy proved NAFLD patients will be recruited in this study for 2 years follow-up. Patients will be assessed at baseline, at every six months for blood count, liver function test, fasting blood-glucose, fasting insulin, ferritin, liver ultrasonography, and liver stiffness.

DETAILED DESCRIPTION:
No.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-70 years of age, 2. liver biopsy proven non alcoholic fatty liver disease. 3. Agree to be followed up regularly; 4. Signature of written informed consent.

Exclusion Criteria:

* 1. Patients with other liver diseases including viral hepatitis, alcoholic liver diseases, autoimmune liver diseases, drug induced liver diseases, genetic metabolic liver disease.

  2. Patients undergone bariatric surgery. 3. HIV infected patients. 4. Pregnant women. 5. Patients with severe diseases with expected survival less than 2 years. 6. Patients had followings before liver biopsy:
  1. Hepatocellular carcinoma or suspected liver cancer,
  2. Decompensated cirrhosis: including ascites, hepatic encephalopathy, esophageal varices bleeding or other complications of decompensated cirrhosis or hepatocelluar carcinoma;
  3. Other malignancy,
  4. Undergone liver transplantation surgery. 7.Patients with any other reasons not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non alcoholic fatty liver disease patients diagnosed with liver biopsy.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-08-23 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
fibrosis progrssion | 2 years
  dynamic changes in liver stiffness measured by VCTE/MRE
steatosis progression | 2 years
  dynamic changes in liver fat measured by controlled attenuation parameter/MRI-PDFF

SECONDARY OUTCOMES:
liver related events | 2 years
  liver decompensation (ascites, variceal bleeding, HE), HCC, liver transplantation, liver relted death.

CONTACTS AND LOCATIONS:
Overall Officials: Hong You, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided